CLINICAL TRIAL: NCT02929004
Title: Chronic Effects of Local Vibration on Neuromuscular Reconditioning After Anterior Cruciate Ligament Reconstruction
Acronym: VIB_LCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1608114; 2016-A01358-43 (Other: ANSM)
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior Cruciate Ligament Reconstruction; Local vibration training; Ligamentoplasty; Anterior cruciate ligament; Corticospinal excitability; Elastography; Knee extensor muscles; Readaptation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibrasens (Experimental): In addition of classical physiotherapist sessions for the readaptation following anterior cruciate ligament reconstruction, this group will follow a local vibration training, using small and portable vibrator device.
  Training programme: vibration training 3/week from Day 1 to Day 60
  Interventions: Device: Vibrasens
- Usual activities (No Intervention): Usual activities from day 1 to Day 60 during their classical physiotherapist sessions for the readaptation following anterior cruciate ligament reconstruction.

INTERVENTIONS:
Device: Vibrasens — Transcutaneous vibrations are used. This device allows vibrations from 25 to 150 Hz with an amplitude of 1 mm. In our study the frequency used is 50 Hz.
  Other Names: Vibrasens (TECHNO CONCEPT, France).
  Arms: Vibrasens

SUMMARY:
These last years, it has been proven that the solicitation of a muscle using vibration may lead to positive effects on the neuromuscular function. Thus, the aim of the current study is to assess if the addition of local vibration training sessions on the quadriceps muscle to the classic readaptation program (i.e. physiotherapist sessions) may allow a better recuperation 2 months after the surgery and the reconstruction of the anterior cruciate ligament.

The aim of the vibration training proposed in the current study is to allow a better recuperation 2 months after the anterior cruciate ligament reconstruction when compared with conventional physiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing to surgery (i.e. ligamentoplasty) of the anterior cruciate ligament

Exclusion Criteria:

* Taking neuro-active substances which can lead to alteration of the corticospinal excitability
* Contra indications for using magnetic stimulation
* Participating in another study in the same time

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary force | 60 days
  Maximal voluntary strength in dorsal flexion of the ankle

SECONDARY OUTCOMES:
6 minutes walking test | 60 days
  The patients will have to realize round trips by walking on a distance of 30 meters during 6 minutes. The total distance traveled by the patient will be calculated (in meters)
Get up and Go test | 60 days
  The patient, sat on a seat placed in 3 meters of the wall, is invited:
  * to get up
  * to walk up to the wall
  * to turn back
  * to return up to their seat and
  * to sit down there again The results will be expressed according to a highly-rated scale from 1 to 5
The cortical level of activation (%) | 60 days
  It is determined by the increment of strength obtained further to a magnetic cortical stimulation realized during a condition of muscle in state of maximal contraction

CONTACTS AND LOCATIONS:
Overall Officials: Pascal EDOUARD, MD, Principal Investigator — CHU de SAINT-ETIENNE; Thomas LAPOLE, PhD, Study Chair — Jean Monnet University
Locations (2):
- France (2):
  - CEPART, Challes-les-Eaux
  - CHU de SAINT-ETIENNE, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coulondre C, Souron R, Rambaud A, Dalmais E, Espeit L, Neri T, Pinaroli A, Estour G, Millet GY, Rupp T, Feasson L, Edouard P, Lapole T. Local vibration training improves the recovery of quadriceps strength in early rehabilitation after anterior cruciate ligament reconstruction: A feasibility randomised controlled trial. Ann Phys Rehabil Med. 2022 Jun;65(4):101441. doi: 10.1016/j.rehab.2020.08.005. Epub 2021 Nov 13. PMID 33059096